CLINICAL TRIAL: NCT06353581
Title: A Phase II Open Label Study of the Efficacy and Safety of Neulapeg (Pegteograstim) in Patients With Locally Advanced or Metastatic Pancreatic Cancer Treated With Modified FOLFIRINOX
Brief Title: Prophylactic Administration of Neulapeg (Pegteograstim) in Patients With Locally Advanced or Metastatic Pancreatic Cancer Receiving the Modified FOLFIRINOX
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 4-2021-0924
Record Dates: First submitted 2024-03-13; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-03

CONDITIONS: Locally Advanced Pancreatic Cancer; Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neulapeg (Experimental): Neulapeg
  Interventions: Drug: Neulapeg; Other: Control
- Control (No Intervention): If grade 3-4 neutropenia or neutropenic fever occurs, patients will be crossover to Neulapeg.

INTERVENTIONS:
Drug: Neulapeg — Participants will receive Neulapeg subcutaneously 24 hours after the end of modified FOLFIRINOX dosing. (Must be administered within a maximum of 72 hours; Neulapeg will only be given for up to 8 cycles).
  Arms: Neulapeg
Other: Control — Patients assigned to the non-Neulapeg arm will be crossover to Neulapeg if they develop grade 3-4 neutropenia or neutropenic fever. Crossover subjects will receive up to 8 cycles of Neulapeg as a secondary treatment regardless of starting cycle.
  Arms: Neulapeg

SUMMARY:
Neutropenia, a decrease in the number of neutrophils, a type of white blood cell, due to the myelosuppressive effects of chemotherapeutic drugs, is a frequent occurrence in patients receiving anticancer drug therapy, which increases the risk of infection, which can have serious consequences such as antibiotic treatment, hospitalization, intensive care unit treatment, and death, and also reduces the effectiveness of anticancer treatment due to dose reduction and cycle delay. Therefore,G-CSF,which acts as a neutrophil growth factor, can be administered immediately after chemotherapy to increase the production rate of neutrophils and promote the efflux of mature neutrophils from the bone marrow, thereby increasing the absolute neutrophil count. Guidelines for the use of G-CSF published by the NCCN indicate that primary prophylaxis with G-CSF has clinical benefit for patients receiving anticancer drug therapy with a risk of febrile neutropenia greater than 20%. For those at 10-20% risk, consider primary prophylaxis based on risk factors. The frequency of neutropenic fever with FOLFIRINOX chemotherapy, which is commonly used in patients with locally advanced or metastatic pancreatic cancer, was 5.4% in a prospective study of patients receiving high-dose regimens, but 42.5% of patients received prophylactic G-CSF, and 63.0% of patients received prophylactic G-CSF compared to 3.0% when given as postoperative adjuvant therapy demonstrating the need for G-CSF administration.In a retrospective study in Japan, a modified FOLFIRINOX chemotherapy regimen without pegylated G-CSF was associated with a 23% incidence of neutropenic fever and 61.5% grade 3-4 neutropenia, while prophylactic administration of pegylated G-CSF was associated with zero neutropenic fever and grade 3-4 neutropenia and longer survival .A retrospective study from Korea also reported that prophylactic G-CSF administration reduced neutropenic fever from 18.5% to 1.8% and Grade 3-4 neutropenia from 55.6% to 31.6 in pancreatic cancer patients receiving FOLFIRINOX .Pegteograstim (Neulapeg®) is a pegylated human recombinant granulocyte colony-stimulating factor with a long half-life (15-80 hours) compared to filgrastim (3-4 hours). Although several studies have demonstrated that G-CSF primary prophylaxis reduces the frequency of hematologic toxicities, particularly febrile neutropenia, during chemotherapy, it has not been prospectively studied whether primary prophylaxis reduces the frequency of grade 3-4 neutropenia and neutropenic fever in the modified FOLFIRINOX chemotherapy regimen in patients with pancreatic cancer. Therefore, this study is designed to determine if prophylactic administration of NEURAPEC reduces the frequency of Grade 3-4 neutropenia and neutropenic fever in patients with locally advanced or metastatic pancreatic cancer receiving modified FOLFIRINOX chemotherapy.

DETAILED DESCRIPTION:
1. Subjects who meet the inclusion/exclusion criteria for this study will be randomized to two arms, Arm A and Arm B, alternating between patients receiving prophylactic Neulapeg and patients not receiving prophylactic Neulapeg. Once assigned, they will be followed until the end of the 8th cycle of modified FOLFIRINOX.
2. Patients assigned to the arm receiving prophylactic Neulapeg will receive Neulapeg subcutaneously 24 hours after the end of modified FOLFIRINOX dosing. (This should be administered no later than 72 hours, and Neulapeg will only be given for a maximum of 8 cycles.)
3. Patients in both arms will have additional visits at the discretion of the investigator for hematologic toxicity surveillance on days 7-10 of modified FOLFIRINOX dosing during the first 4 cycles. Thereafter, patients will be seen only at the time of chemotherapy administration at the discretion of the investigator.
4. Patients in both arms will be instructed to return for any fever greater than 38.3 degrees Celsius or greater than 38.0 degrees Celsius lasting more than 1 hour.
5. Patients assigned to the arm not receiving prophylactic Neulapeg will not receive intervention with G-CSF for neutropenia of grade 2 or less.
6. Patients assigned to the no prophylactic Neulapeg arm will be crossover to prophylactic Neulapeg if they develop Grade 3-4 neutropenia or neutropenic fever. Crossover subjects will receive up to 8 cycles of prophylactic Neulapeg as a secondary treatment regardless of starting cycle.
7. Hematologic toxicity monitored every cycle for 8 cycles / Quality of life assessed according to EORTC QLQ-C30 at baseline, once every 2 weeks for a total of 5 times (Baseline, Cycle 2 Day 1, Cycle 4 Day1 , Cycle 6 Day 1 , Cycle 8 Day 1) / completion of the bone pain questionnaire at baseline, once every 1 cycle for the first 4 cycles, and then every 2 cycles for a total of 7 times (Baseline, Cycle 1 Day 1, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 6 Day 1, Cycle 8 Day 1). The mFOLFIRINOX will be administered every 2 weeks for up to 8 cycles, while Neulapeg will be administered within 24-72 hours of the end of dosing and will be available for up to 8 cycles only. The crossover control arm will continue as usual.
8. The modified FOLFIRINOX chemotherapy regimen will be administered at the original dose at the start of Cycle 1, with subsequent dose deferral until recovery of a neutrophil count ≥1,000 /mm3 in the event of toxicity, with dose reduction at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pancreatic cancer assessed as locally advanced or metastatic by histology/cytology or imaging studies including CT or MRI
2. Patients who are scheduled to receive modified FOLFIRINOX chemotherapy (less than second-line treatment as a consolidation regimen)
3. Patients with an ECOG performance capacity index of 0 to 1
4. Patients 19 years of age or older who are willing and able to complete a written informed consent for this study
5. Patients with adequate organ function
6. Patients who voluntarily agree to participate in the study

Exclusion Criteria:

1. Other histologic/cytologic or imaging diagnosis other than pancreatic ductal adenocarcinoma (e.g., neuroendocrine tumor, etc.)
2. Patients with moderate acute or chronic medical conditions or abnormal laboratory findings that would affect the results of this study.
3. Pregnant or lactating women or patients planning to become a mother during the scheduled study period from the screening visit through Day 120 after the last dose of study drug
4. Active systemic infection that is not resolving

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2024-05-08 (Estimated); Study Completion 2024-05-08 (Estimated)

PRIMARY OUTCOMES:
Development of grade 3-4 neutropenia (grade 3-4 neutropenia, ANC<1000/mL) | 4 years
  The occurrence of grade 3-4 neutropenia (grade 3-4 neutropenia, ANC<1000/mL) and the occurrence of neutropenic fever (febrile neutropenia) will be tested using the chi-squared test.
development of neutropenic fever (febrile neutropenia) | 4 years
  The occurrence of grade 3-4 neutropenia (grade 3-4 neutropenia, ANC<1000/mL) and the occurrence of neutropenic fever (febrile neutropenia) will be tested using the chi-squared test.

SECONDARY OUTCOMES:
relative dose intensity | 4 years
  Relative dose intensity: proportion of administrated dose per m2 of BSA per week in relation to optimal dose per m2 of BSA per week
quality of life assessed according to EORTC QLQ-C30 | 4 years
  The EORTC QLQ-C30 assesses health-related quality of life in cancer patients participating in clinical trials. The EORTC QLQ-C30 comprises 5 functional scales (physical, role, emotional, social, cognitive), 8 single-item symptom scales (fatigue, pain, nausea/vomiting, appetite loss, constipation, diarrhea, insomnia, and dyspnea), as well as subscales assessing global health/quality of life and financial impact. Raw scores are transformed to a scale of 0 to 100, with higher scores representing better functioning/quality of life and greater symptom burden.
Number of patients experiencing Adverse events (AEs) | 4 years
  An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention whether or not considered related to the study intervention.
objective response rate | 4 years
  Objective response rate is defined as the proportion of participants with a complete response (CR) or partial response (PR) based on RECIST v1.1
Progression-free survival | 4 years
  Progression-free survival is defined as the time from randomization to the first occurrence of radiographic progression based on RECIST version 1.1 per investigator or death from any cause.
Overall survival | 4 years
  Overall survival is defined as the time from randomization to the event of death from any cause.
Change in blood cytokine concentrations | 4 years
  Changes in blood cytokine concentrations: measured by ELISA, tested by t-test G-CSF induced bone pain assessed by questionnaire G-CSF induced bone pain modality, assessed by questionnaire, will be measured by the area under the curve (AUC) of the pain scores recorded by the patients. objective response rate according to CTCAE v5.0 will be tested using the chi-squared test will be used to test for differences in adverse events and objective response rates according to CTCAE v5.0.
  Differences in progression-free survival, overall survival, and progression-free survival will be analyzed using the Kaplan-Meier test. (overall survival) .Questionnaire-based endpoints such as QOL will be assessed up to Week 8. QOL and other survey-based endpoints will continue to be administered up to cycle 8, and survival will only be validated in patients who did non-crossover
G-CSF induced bone pain as assessed by questionnaires | 4 years
  G-CSF induced bone pain assessed by questionnaire G-CSF induced bone pain modality, assessed by questionnaire, will be measured by the area under the curve (AUC) of the pain scores recorded by the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee CK, Kim I, Seo DH, Park S, Kim M, Lee SH, Lee YJ, Kim JH, Kim CG, Choi HJ. Pegylated granulocyte colony-stimulating factor primary prophylaxis versus no prophylaxis in patients with unresectable pancreatic cancer treated with modified-FOLFIRINOX: a randomized, open-label, multicenter, phase 2 trial. EClinicalMedicine. 2025 Nov 14;90:103646. doi: 10.1016/j.eclinm.2025.103646. eCollection 2025 Dec. PMID 41324016